CLINICAL TRIAL: NCT06532058
Title: Safety and Efficacy of QHRD107 Capsule Combined With Venclexta and Azacitidine in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia: a Single-arm, Open, Multicenter Phase IIa Study
Brief Title: Phase IIa Study to Assess Safety and Efficacy in the Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changzhou Qianhong Bio-pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QH-RD107-02-01
Record Dates: First submitted 2024-07-20; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (R/R-AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: a single-arm, open, multicenter Phase IIa study with dose escalation and dose extension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part-A (Cohort 1-3) (Experimental): Three dose groups were set up. The doses of QHRD107 capsules were 40 mg Q12H, 60 mg Q12H and 80 mg Q12H, respectively, combined with Venclexta and Azacitidine.
  Interventions: Drug: QHRD107 capsule，Venclexta and Azacitidine
- Part-B (Cohort 1-2) (Experimental): Cohort 1： [QHRD107 capsule 60mg Q12H D1-28]+[Venclexta QD D1-28]+[Azacitidine QD D1-7]; Cohort 1：[QHRD107 capsule 80mg Q12H D1-28]+[Venclexta QD D1-28]+[Azacitidine QD D1-7] .
  Interventions: Drug: QHRD107 capsule，Venclexta and Azacitidine

INTERVENTIONS:
Drug: QHRD107 capsule，Venclexta and Azacitidine — QHRD107（orally），Venclexta（orally），Azacitidine（subcutaneous injection）
  Other Names: CDK9 inhibitors

SUMMARY:
The purpose of this study is to assess the safety and efficacy of QHRD107 capsule combined with Venclexta and azacitidine in the treatment of relapsed/refractory acute myeloid leukemia: a single-arm, open, multicenter Phase IIa study

DETAILED DESCRIPTION:
This study is a single-arm, open, multicenter phase IIa clinical study, which is divided into two stages: the dose-increasing study phase and the dose-expanding exploration phase. The purpose of the dose-escalation phase is to explore the safety and tolerability of QHRD107 capsule（40mgBID,60mgBID and 80mgBID） combined with Venclexta and azacitidine, to evaluate the efficacy of the three-drug combination in subjects with relapsed/refractory acute myeloid leukemia (R/R-AML), and to explore the pharmacokinetic characteristics of the combination. The dose expansion stage aims to further evaluate the safety, efficacy, pharmacodynamics and pharmacokinetics of QHRD107 capsule（60mgBID and 80mgBID）combined with Venclexta and azacitidine on the basis of exploring the safe dose range determined in the dose escalation stage, and determine the recommended dose for subsequent clinical studies

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign informed consent;
2. Age 18 and above;
3. Subjects with confirmed International Consensus Classification (ICC) relapsed/refractory acute myeloid leukemia (R/R-AML) :

   Recurrence was defined as the recurrence of leukemia cells in peripheral blood or ≥5% of bone marrow original cells after complete response (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or the occurrence of extramedullary leukemia cell infiltration.

   Refractory is defined as meeting any of the following criteria:
   1. Initial treatment cases that failed after 2 courses of treatment with standard protocols;
   2. Relapse within 12 months after complete remission (CR) after consolidation and intensive treatment;
   3. Recurrence after 12 months but failed to respond to conventional chemotherapy;
   4. Two or more relapses.
4. ECOG evaluation ≤2 points;
5. Expected survival ≥3 months;
6. White blood cell (WBC) count <25×109 cells /L (hydroxyurea is allowed to control the white blood cell count before treatment);
7. Subjects must have adequate liver function: total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN;
8. Subjects must have adequate renal function: creatinine clearance ≥50 mL/min (calculated using the Cockroft-Gault formula);
9. The subject has recovered from previous therapeutic toxicity to < grade 2 (according to CTCAE 5.0 criteria), excluding primary disease effects. The following are excluded: hair loss, fatigue, hyperpigmentation, stable hypothyroidism with hormone replacement therapy, peripheral nerve toxicity after chemotherapy;
10. Eluting period from the first administration of antitumor therapy: a) At least 2 weeks between the end of cytotoxic chemotherapy drug treatment; b) Non-cytotoxic drugs should be separated by at least 5 half-lives (if the duration of 5 half-lives exceeds 4 weeks, the washout period is still measured by 4 weeks), and the interval > 4 weeks shall prevail if the half-life is not clear; c) Anti-tumor Chinese medicine at least 2 weeks interval;
11. Ability to understand and conduct visits, treatments, laboratory tests, and other research procedures as planned;
12. Male/female subjects with reproductive potential must use effective contraception from the date of signing the informed consent until 6 months after the last trial medication. At the same time, male subjects with reproductive potential must refrain from sperm donation from signing their informed consent until six months after the last trial medication.

Exclusion Criteria:

1. Subjects previously treated with other CDK9 inhibitors;
2. Subjects who are allergic to the active ingredients and/or excipients of the investigational drugs (QHRD107, Veneckla, and azacytidine);
3. Subjects with a history of myeloproliferative tumors (MPN);
4. Subjects with a history of chronic myeloid leukemia (CML);
5. Subjects with Ph chromosome-positive or BCR-ABL fusion gene positive acute myeloid leukemia (AML);
6. Confirmed acute promyelocytic leukemia;
7. Patients with AML central nervous system infiltration;
8. Subjects with extramedullary leukemia (such as myeloid sarcoma, skin infiltration, etc.) (except extramedullary lesions such as liver, spleen, and lymph node involvement);
9. Human immunodeficiency virus (HIV) antibody positive subjects; Subjects with active HBV infection: hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive, and peripheral blood hepatitis B virus (HBV-DNA) higher than the upper limit of normal; Subjects with active HCV infection: HCV antibody positive, peripheral blood HCV RNA positive;
10. The subject has an active infection (including bacterial, viral, and fungal infections) that requires systemic antibiotic treatment as determined by the investigator to be clinically significant;
11. People with significant active cardiovascular disease within the previous 6 months, including but not limited to: ≥III Heart failure as defined by the New York Heart Association (NYHA); Angina pectoris requiring surgical treatment, unstable angina pectoris, myocardial infarction; Hypertension that remains poorly controlled after treatment (i.e., systolic ≥160 mmHg, diastolic ≥90 mmHg); Uncontrolled arrhythmias; The left ventricular function resting ejection fraction measured by echocardiography was less than 50%. QT interval: > 450 ms for men and > 470 ms for women (according to the QTcF formula), or are on medication known to lengthen the QT/QTc interval, or have other factors that may lengthen the QTc interval; Or for patients whose QT interval is still > 450 ms after QT interval prolongation treatment;
12. Patients who have received allogeneic hematopoietic stem cell transplantation within 60 days of their initial investigational treatment must discontinue all immunosuppressants during the investigational treatment;
13. Patients who have previously received CAR-T therapy;
14. The subject has a malabsorption syndrome or other comorbid condition that prevents him from swallowing the capsule or administering the drug through enteral channels;
15. A history of other malignancies in the past 5 years, excluding cured basal cell carcinoma of the skin, localized squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or carcinoma in situ of the breast;
16. Pregnant or lactating women, or subjects who are fertile and do not want to take effective contraceptive measures;
17. Any ill-controlled clinical problems (such as severe psychiatric, neurological, cardiovascular, respiratory, digestive, urinary, etc.) or other factors that the investigator believes prevented the subject from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose（Dose Escalation Phase） | From screenng through to 28 day follow up period
  Enrolled subjects performed dose climbing according to the "3+3 principle".The highest dose of DLT（Dose-Limiting Toxicity） incidence 1/6 is MTD
The Compound complete response rate (CCR) and the corresponding mitigation duration (DORccr)（Dose expansion phase） | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  The Compound complete response rate (CCR) was defined as the percentage of participants who achieved complete remission(CR),CR with partial hematologic recovery(CRh),CR with incomplete hematologic recovery (CRi) per the European LeukemiaNet (ELN) recommendations for AML. CR was defined as bone marrow blasts < 5%, absence of circulating blasts,absence of extramedullary disease,ANC ≥ 1.0 × 10˄9/L (1,000/µL),platelet count ≥ 100 × 10˄9/L (100 000/µL).CRh was defined as ANC ≥ 0.5 × 10˄9/L (500/µL) and platelet count ≥ 50 × 10˄9/L (50000/µL), otherwise all other CR criteria met.CRi was defined as all CR criteria except for residual neutropenia < 1.0 × 10˄9/L (1,000/µL) or thrombocytopenia < 100 × 10˄9/L (100 000/µL).DORccr refers to the time between the first assessment of efficacy reaching CR/CRi/CRh/MLFS/PR and the first assessment of disease recurrence or death from any cause.

SECONDARY OUTCOMES:
Safety as assessed by incidence ,severity,and causality of adverse events | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  The frequency and number of Adverse events
Plasma measurements of QHRD107 | At the end of Cycle 1 (each cycle is 28 days)
  The concentration of QHRD107 was measured at 3 different doses
Complete Remission Rate | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  The complete remission (CR) rate was defined as the percentage of participants who achieved CR per the ELN criteria for AML.
Objective Remission Rate | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  The objective remission rate (ORR) was defined as the percentage of participants who achieved CR, CRh, CRi,morphologic leukemia-free state (MLFS),or partial remission (PR) per the ELN for AML.Partial remission (PR) was defined as normalization in peripheral blood neutrophil and platelet counts with at least a 50% decrease in blasts persisting in bone marrow versus baseline.MLFS was defined as bone marrow blasts < 5%,absence of circulating blasts, absence of extramedullary disease, no hematologic recovery required.
Duration of Remission(DOR) | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  Duration of remission was defined as the number of days from the date of first remission (CR, CRi, or PR) per the IELN criteria for AML to the earliest recurrence or progressive disease (PD).
Time to first CR, CRi, CRh,MLFS,and PR | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  Time to first CR, CRi, CRh,MLFS,and PR was defined as the time from the start of the first dose until the first observation of CR or CRh or CRi or MLFS or PR
Rate of Minimal Residual Disease (MRD) Negativity | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  The rate of minimal residual disease (MRD) response was defined as the percentage of participants who had MRD negative status.
Event-free lifetime | From the date of the patient first received treatment to the end of the fourth cycle（each cycle is 28 days）
  For all subjects, the time from first dosing to treatment failure, or disease recurrence, or death from any cause, whichever occurred first. Treatment ineffectiveness was defined as failure to achieve CR, CRh, CRi, or MLFS after ≤4 cycles of treatment.
Overall survival | 1 year
  Overall survival(OS) was defined as the time from the date of first treatment to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Li Junmin, Doctor, Principal Investigator — Ruijin Hospital
Locations (10):
- China (10):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Huai 'an First People's Hospital, Huaian, Jiangsu
  - Zhongda Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - ShengJing Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - Tongren Hospital Shanghai Jiao Tong University School Of Medicine, Shanghai, Shanghai Municipality
  - Ruijin hospitol, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No